CLINICAL TRIAL: NCT05702333
Title: Postoperative Prolonged Vasoactive-inotropic Support and Levosimendan Use After Lung Transplantation: a Retrospective Analysis of Risk Factors and Impact on Outcomes
Brief Title: Vasoactive-inotropic Support and Levosimendan Use After Lung Transplantation
Acronym: VASO_LUTX
Status: Completed | Type: Observational
Sponsor: Policlinico Hospital (Other)
Responsible Party: Principal Investigator, Giacomo Grasselli, Prof., Policlinico Hospital
Other Study IDs: VASO_LUTX
Record Dates: First submitted 2023-01-18; First posted 2023-01-27 (Actual); Last update posted 2023-04-05 (Actual); Status verified 2023-04

CONDITIONS: Lung Transplant; Complications
Keywords: Lung Transplant; Vasoactive drugs

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Vasoactive-inotropic drug use (VASO+): All patients treated with vasoactive-inotropic drugs (epinephrine, norepinephrine, dobutamine, dopamine, and levosimendan) after 12 hours after Intensive Care Unit Admission were retrospectively classified in the VASO + cohort.
  Interventions: Drug: Epinephrine Norepinephrine Dobutamine Dopamine Levosimendan
- No vasoactive-inotropic drug (VASO -): Patients treated with vasoactive-inotropic drugs (epinephrine, norepinephrine, dobutamine, dopamine, and levosimendan) in the first 12 hours after Intensive Care Unit Admission (ICU) or patients never treated with such drugs in ICU were retrospectively classified in the VASO - cohort.

INTERVENTIONS:
Drug: Epinephrine Norepinephrine Dobutamine Dopamine Levosimendan — Vasoactive-inotropic drugs were administered according to clinical decision of the doctor in charge.
  Groups: Vasoactive-inotropic drug use (VASO+)

SUMMARY:
Bilateral Lung transplantation (LUTX) is performed in selected patients with end-stage respiratory failure. During surgery, pulmonary arteries are sequentially cross-clamped. This can cause acute heart failure and hemodynamic instability that eventually persist into the postoperative period, leading to the need for prolonged vasoactive support in the postoperative Intensive Care Unit. Levosimendan is a relatively new vasoactive-inotropic drug, with different pharmacodynamic properties.

This observational retrospective cohort study primarily aims 1) to describe the need for prolonged vasoactive support; 2) to evaluate the risk factors for prolonged vasoactive support; 3) to assess the impact of prolonged vasoactive support on outcomes. The secondary aim is to describe the use of Levosimendan in this cohort of patients.

ELIGIBILITY:
Inclusion Criteria:

Intensive Care Unit admission after Double Lung Transplant surgery.

Exclusion Criteria:

1. single Lung Transplantation;
2. re-transplantation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: We retrospective enrolled all consecutive patients admitted to ICU after bilateral lung transplantation from February 2017 to July 2022.
Sampling Method: Non-Probability Sample
Enrollment: 150 (Actual)
Dates: Start 2017-02-01 (Actual); Primary Completion 2022-07-31 (Actual); Study Completion 2022-07-31 (Actual)

PRIMARY OUTCOMES:
Need of postoperative vasoactive support after LUTX | February 2017 - July 2022
  This outcome aims to describe the number of patients treated with vasoactive drugs after Lung Transplantation in Intensive Care Unit, and median dosage and duration of therapy.
Postoperative vasoactive support use after LUTX risk factors. | February 2017 - July 2022
  This outcome aims to assess if preoperative characteristics or intraoperative events can represent risk or protecting factors for postoperative vasoactive drugs need.
Vasoactive support after LUTX impacts on outcomes. | February 2017 - July 2022
  This outcome aims to assess if the vasoactive drug use in the postoperative management of Lung Transplanted patients impacts 1) mechanical ventilation duration; 2) Continuous Renal Replacement Therapy; 3) ICU and Hospital Length of Stay; 4) Primary Graft Dysfunction; 5) in-hospital mortality; 6) survival at July 31st, 2023.

SECONDARY OUTCOMES:
Description of Levosimendan use in post-operative LUTX patients. | February 2017 - July 2022
  This outcome aims to describe the number and the characteristics of patients treated with levosimendan.

CONTACTS AND LOCATIONS:
Overall Officials: Vittorio Scaravilli, MD, Principal Investigator — University of Milan
Locations (1):
- Fondazione IRCCS Ca'Granda - Ospedale Maggiore Policlinico, Milan, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Mal H, Dehoux M, Sleiman C, Boczkowski J, Leseche G, Pariente R, Fournier M. Early release of proinflammatory cytokines after lung transplantation. Chest. 1998 Mar;113(3):645-51. doi: 10.1378/chest.113.3.645. PMID 9515837
- [Background] Di Nardo M, Tikkanen J, Husain S, Singer LG, Cypel M, Ferguson ND, Keshavjee S, Del Sorbo L. Postoperative Management of Lung Transplant Recipients in the Intensive Care Unit. Anesthesiology. 2022 Mar 1;136(3):482-499. doi: 10.1097/ALN.0000000000004054. PMID 34910811
- [Background] Todd TR. Early postoperative management following lung transplantation. Clin Chest Med. 1990 Jun;11(2):259-67. PMID 2189661
- [Background] Guillen RV, Briones FR, Marin PM, Jover AS, Represa JM, Colom AP. Lung graft dysfunction in the early postoperative period after lung and heart lung transplantation. Transplant Proc. 2005 Nov;37(9):3994-5. doi: 10.1016/j.transproceed.2005.09.193. PMID 16386607